CLINICAL TRIAL: NCT00005557
Title: Epidemiology of Sleep-Disordered Breathing in Adults
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0084; R01HL062252 (NIH); A538500 (Other: UW, Madison); SMPH/POP HEALTH SCI/POP HLTH (Other: UW, Madison)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Sleep Disorders; Cerebrovascular Disorders; Cardiovascular Disease; Neurologic Disorders; Mood Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Cerebrovascular Disorders; Cardiovascular Diseases; Nervous System Diseases; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize the natural history and biologic spectrum of sleep disordered breathing (SDB) and other sleep problems and disorders, and test hypotheses regarding the causes and consequences of SDB and other sleep problems and disorders.

DETAILED DESCRIPTION:
BACKGROUND:

Recent research has shown that sleep disordered breathing (SDB) is much more common than previously thought. While it is known that in clinic samples, SDB is associated with hypertension, cardiovascular disease and mortality, little is known about the natural history of this disorder, particularly in the general population, nor about the causal role of known risk factors. The knowledge obtained from the results of this study will help advance the field of sleep disorders medicine. Information about longitudinal effects and causal relationships may be applied to clinical situations, thus reducing the morbidity and mortality associated with this disorder.

DESIGN NARRATIVE:

In this longitudinal study, follow-up polysomnography and other protocols are conducted on an established cohort of men and women (age 30-60 years at the time of initial recruitment in 1989), currently enrolled in the Wisconsin Sleep Cohort Study. The study aims to : 1) describe the natural history of SDB across middle and older age; 2) investigate associations of SDB with early and intermediate markers of cardiovascular dysfunction, damage, and cardiovascular disease; 3) investigate the longitudinal association of SDB in accelerated cognitive decline; 4) investigate the association of SDB and adverse sleep characteristics with age-related risk factors and outcomes.

ELIGIBILITY:
Inclusion criteria:

* Employee of one of the 4 Wisconsin state agencies
* Age 30-60 in 1988

Exclusion criteria:

* Current pregnancy
* Unstable or decompensated cardiopulmonary disease
* Airway cancer
* Recent upper respiratory surgery

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In 1988, employees of 4 Wisconsin state agencies, ages 30-60 years, were surveyed regarding sleep habits and problems by mail. From these data, a sampling frame was constructed and 2884 randomly-selected men and women (of 4896 survey respondents) were invited to participate in the WSC Study. Recruitment for baseline sleep studies occurred from 1989 to 2004.
Sampling Method: Probability Sample
Enrollment: 1545 (Actual)
Dates: Start 1999-04; Primary Completion 2028-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
sleep disorders and problems, cardiovascular and cognitive outcomes | measured at each study visit
  Overnight polysomnography is used to assess sleep pathology. Questionnaires are used to assess sleep habits. A variety of clinical and laboratory assessments measure cardiovascular and cognitive outcomes.

SECONDARY OUTCOMES:
cardiovascular outcomes | measured at each study visit
  A variety of clinical and laboratory assessments measure cardiovascular outcomes.

OTHER OUTCOMES:
cognitive outcomes | measured at each study visit
  A variety of clinical and laboratory assessments measure cognitive outcomes.
gait and balance | measured at each study visit
  A series of walking tests are conducted.
mental health outcomes | evaluated at each study visit
  Questionnaires assess mood, depression, and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Peppard, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Peppard PE, Young T, Palta M, Dempsey J, Skatrud J. Longitudinal study of moderate weight change and sleep-disordered breathing. JAMA. 2000 Dec 20;284(23):3015-21. doi: 10.1001/jama.284.23.3015. PMID 11122588
- [Background] Young T, Finn L, Palta M. Chronic nasal congestion at night is a risk factor for snoring in a population-based cohort study. Arch Intern Med. 2001 Jun 25;161(12):1514-9. doi: 10.1001/archinte.161.12.1514. PMID 11427099
- [Background] Kadotani H, Kadotani T, Young T, Peppard PE, Finn L, Colrain IM, Murphy GM Jr, Mignot E. Association between apolipoprotein E epsilon4 and sleep-disordered breathing in adults. JAMA. 2001 Jun 13;285(22):2888-90. doi: 10.1001/jama.285.22.2888. PMID 11401610
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Punjabi NM, Bandeen-Roche K, Young T. Predictors of objective sleep tendency in the general population. Sleep. 2003 Sep;26(6):678-83. doi: 10.1093/sleep/26.6.678. PMID 14572120
- [Background] Young T, Rabago D, Zgierska A, Austin D, Laurel F. Objective and subjective sleep quality in premenopausal, perimenopausal, and postmenopausal women in the Wisconsin Sleep Cohort Study. Sleep. 2003 Sep;26(6):667-72. doi: 10.1093/sleep/26.6.667. PMID 14572118
- [Background] Lin L, Finn L, Zhang J, Young T, Mignot E. Angiotensin-converting enzyme, sleep-disordered breathing, and hypertension. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1349-53. doi: 10.1164/rccm.200405-616OC. Epub 2004 Sep 24. PMID 15447944
- [Background] Peppard PE, Young T. Exercise and sleep-disordered breathing: an association independent of body habitus. Sleep. 2004 May 1;27(3):480-4. doi: 10.1093/sleep/27.3.480. PMID 15164902
- [Background] Reichmuth KJ, Austin D, Skatrud JB, Young T. Association of sleep apnea and type II diabetes: a population-based study. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1590-5. doi: 10.1164/rccm.200504-637OC. Epub 2005 Sep 28. PMID 16192452
- [Background] Arzt M, Young T, Finn L, Skatrud JB, Bradley TD. Association of sleep-disordered breathing and the occurrence of stroke. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1447-51. doi: 10.1164/rccm.200505-702OC. Epub 2005 Sep 1. PMID 16141444
- [Derived] Kuo WC, Bratzke LC, Hagen EW, Hale L, Brown RL, Barnet JH, Peppard PE. Metabolic health disparities driven by financial stress: Behavioural adaptation or modification? Stress Health. 2023 Aug;39(3):614-626. doi: 10.1002/smi.3210. Epub 2022 Dec 1. PMID 36413205
- [Derived] Kuo WC, Ersig AL, Johnson HM, Brown RL, Oakley LD, Hagen EW, Barnet JH, Peppard PE. Association between stressful life events and non-optimal lipid levels among women with hyperlipidaemia. Eur J Cardiovasc Nurs. 2023 Mar 1;22(2):210-219. doi: 10.1093/eurjcn/zvac032. PMID 35714051
- [Derived] Kuo WC, Oakley LD, Brown RL, Hagen EW, Barnet JH, Peppard PE, Bratzke LC. Gender Differences in the Relationship Between Financial Stress and Metabolic Abnormalities. Nurs Res. 2021 Mar-Apr 01;70(2):123-131. doi: 10.1097/NNR.0000000000000489. PMID 33630535